CLINICAL TRIAL: NCT00563862
Title: Prospective Randomized Study on Therapeutic Gain Achieved By Chemoradiation And/Or Accelerated Radiation For T3-4N0-1M0 Nasopharyngeal Carcinoma
Brief Title: Benefit of Adding Chemotherapy And/Or Modification of Radiotherapy Schedule for Advance Nasopharyngeal Carcinoma (T3-4N0-1M0)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The Hong Kong Nasopharyngeal Cancer Study Group (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: L/M-78 to PYH 08/79; HARECCTR0500024; NPC99-02
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Nasopharyngeal Neoplasms; Carcinoma, Squamous Cell
Keywords: Nasopharyngeal Carcinoma; T3-4N0-1M0
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Carcinoma, Squamous Cell; Nasopharyngeal Carcinoma | interventions — Cisplatin; Fluorouracil

INTERVENTIONS:
Procedure: Conventional RT
Procedure: Accelerated RT
Drug: Cisplatin
Drug: 5-fluorouracil

SUMMARY:
To test the therapeutic ratio of accelerated radiotherapy and/or chemotherapy on locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Undifferentiated or non-keratinizing carcinoma
* Tumor staged as T3-4 AND N0-1
* No evidence of distant metastasis (M0)
* Performance status: 0-2
* Marrow: WBC >= 4 and platelet = 100
* Renal: creatinine clearance = 60
* Informed consent

Exclusion Criteria:

* WHO type I squamous cell carcinoma or adenocarcinoma
* Age >= 70
* Palliative intent or tumor extent mandating AP opposing facio-cervical fields
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years
* Previous radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume
* Previous chemotherapy
* Patient is pregnant or lactating

Max Age: 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 1999-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Failure free survival rate | 5-year

SECONDARY OUTCOMES:
Overall survival rate | 5-year
Disease-specific survival rate | 5-year
Complication-free rates | 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Anne WM Lee, Dr, Principal Investigator — Department of Clinical Oncology, Pamela Youde Nethersole Eastern Hospital
Locations (5):
- China (5):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong